CLINICAL TRIAL: NCT02652000
Title: Retrospective Analysis of Quality of Life After Permanent Interstitial Iodine Seed Brachytherapy for Prostate Cancer
Brief Title: Quality of Life After Permanent Interstitial Iodine Seed Prostate Brachytherapy
Status: Completed | Type: Observational
Sponsor: Kantonsspital Graubuenden (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Daniel Rudolf Zwahlen, MD, MBA, Kantonsspital Graubuenden
Other Study IDs: KEK-ZH-Nr. 2015-0573
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasms, Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention in this retrospective study — No Intervention in this retrospective Analysis.

SUMMARY:
Retrospective study to analyze Quality of life in men after iodine seed brachytherapy for localized prostate cancer

DETAILED DESCRIPTION:
Retrospective Evaluation of Quality of life data collected on men who underwent iodine seed brachytherapy at the University Hospital Zurich

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years of age
* iodine seed brachytherapy for localized prostate cancer at the University Hospital Zurich

Exclusion Criteria:

* No iodine seed brachytherapy for localized prostate cancer at the University Hospital Zurich

Ages: 48 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had idodine seed brachytherapy for localized prostate cancer between 2009 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
CTCAE v4.03ff Grade 1-4 Sexual/Reproductive Function | 5 years (2009-2014)
  Scale

SECONDARY OUTCOMES:
CTCAE v4.03ff Grade 1-4 Gastrointestinal | 5 years (2009-2014)
  Scale
CTCAE v4.03ff Grade 1-4 Renal/Genitourinary | 5 years (2009-2014)
  Scale
International Prostate Symptom Score (IPSS) | 5 years (2009-2014)
  Scale
International Index of erectile function, five items (IIEF-5) | 5 years (2009-2014)
  Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Zwahlen, MD, MBA, Principal Investigator — Kantonsspital Graubuenden
Locations (1):
- Kantonsspital Graubuenden, Department of Radiaton Oncology, Chur, Switzerland